CLINICAL TRIAL: NCT05168826
Title: SAPIEN 3 China Post Market Registry Study
Brief Title: China S3 PMS: SAPIEN 3 China Post Market Registry Study
Status: Active, not recruiting | Type: Observational
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Other Study IDs: 2021-06
Record Dates: First submitted 2021-12-10; First posted 2021-12-23 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Aortic Stenosis, Severe
Keywords: Transcatheter aortic valve implantation (TAVI); Transcatheter aortic valve replacement (TAVR); SAPIEN 3; Heart disease; Cardiovascular disease
MeSH Terms: conditions — Aortic Valve Stenosis; Heart Diseases; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Transcatheter Aortic Valve Implantation (TAVI)
  Interventions: Device: SAPIEN 3 Transcatheter Heart Valve

INTERVENTIONS:
Device: SAPIEN 3 Transcatheter Heart Valve — Implantation of the SAPIEN 3 valve

SUMMARY:
The objective of this study is to evaluate the long term safety and effectiveness of the SAPIEN 3 Transcatheter Heart Valve system in real world setting.

DETAILED DESCRIPTION:
This is an observational, single-arm, multicentre, post-market study.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with symptomatic, severe, calcified aortic stenosis who is appropriate for the treatment with transcatheter aortic valve replacement as determined by a heart team and will undergo TAVI with the Edwards SAPIEN 3 System as part of standard-of-care treatment
2. All surgical risks as determined by the site Heart Team
3. The subject or subject's legal representative has been informed of the nature of the study, agrees to its provisions and has provided written informed consent.

Exclusion Criteria:

1. Medical, social, or psychological conditions that preclude appropriate consent and follow-up, including subjects under guardianship
2. Considered to be part of a vulnerable population
3. Pre-existing mechanical or bioprosthetic aortic valve
4. Active SARS-CoV-2 infection or previously diagnosed with COVID-19 with sequelae that could confound endpoint assessments
5. Cannot tolerate an anticoagulation/antiplatelet regimen
6. Evidence of intracardiac mass, thrombus, vegetation, active infection or endocarditis
7. Tortuous or calcified vessels that would prevent safe entry of the dilators and sheath
8. Participating in a drug or device study that has not reached its primary endpoint

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects who will undergo TAVI with the Edwards SAPIEN 3 System.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2022-01-24 (Actual); Primary Completion 2035-12 (Estimated); Study Completion 2035-12 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | 10 years
  The number of patients that died

CONTACTS AND LOCATIONS:
Locations (14):
- China (14):
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Xiamen Cardiovascular Hospital Xiamen University, Xiamen, Fujian
  - First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - Henan Provincial Chest Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Union Hospital Affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Shanghai General Hospital, Shanghai, Shangahi
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality
  - Xinhua Hospital Affiliated to Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital of Xi'an Jiao Tong University, Xi’an, Shanxi
  - First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - People's Hospital of Xinjiang Uygur Autonomous Region, Ürümqi, Xinjiang
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No